CLINICAL TRIAL: NCT04991168
Title: Oral Health and Diabetes: Relationship Between Knowledge, Practices and Oral Health Status in Patients Followed in the Diabetes Department at the Montpellier University Hospital.
Brief Title: Relationship Between Oral Health and Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0504
Record Dates: First submitted 2021-07-27; First posted 2021-08-05 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Diabetes
Keywords: Oral hygiene; Public Health; Patients coming to the CHU Lapeyronie for consultation or those being hospitalised there; Prevention; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients over 18 from the CHU Lapeyronie: Diabetic patients over 18 from the CHU Lapeyronie
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Two questionnaires used to assess the state of knowledge and practices in oral health. An oral assessment will be carried out for voluntary patients.

SUMMARY:
The aim of this study is to assess the state of knowledge and practices in oral health of diabetic patients through the use of two questionnaires. It is also to analyse the link between the oral health status and the profile of diabetic patient, by carrying out an oral assessment for voluntary patients.

ELIGIBILITY:
Inclusion criteria:

- All diabetic patients over 18 coming to the CHU Lapeyronie

Exclusion criteria:

-Non diabetic patients, diabetic patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic patients over 18 coming to the CHU Lapeyronie
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Oral health knowledge and practice questionnaire score. | 1 day
  Oral health knowledge and practice questionnaire score.
Number of missing and decayed teeth on the oral examination and clinical signs in diabetology. | 1 day
  Number of missing and decayed teeth on the oral examination and clinical signs in diabetology.

CONTACTS AND LOCATIONS:
Overall Officials: Camille INQUIMBERT, PhD, Study Director — University Hospital, Montpellier; Amir MEZIANE, resident, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC